CLINICAL TRIAL: NCT07042191
Title: DISCO Provider: A Multi-level Intervention to Reduce Financial Toxicity in Patients With Cancer Through Improved Treatment Cost Discussions
Brief Title: A Provider Intervention to Reduce Financial Toxicity in Patients With Cancer Through Improved Treatment Cost Discussions
Acronym: DISCO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Barbara Ann Karmanos Cancer Institute (Other)
Responsible Party: Principal Investigator, Lauren Hamel, Principal Investigator, Barbara Ann Karmanos Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2022-085
Record Dates: First submitted 2025-05-23; First posted 2025-06-27 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-05

CONDITIONS: Healthy; Financial Toxicity
MeSH Terms: conditions — Financial Stress

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- DISCO (Discussions of Cost) Provider Companion Intervention (Experimental): Providers of Cancer patients at Karmanos Cancer Institute will use the DISCO (Discussion of Cost) provider communication intervention to assess its feasibility, acceptability, and usability
  Interventions: Behavioral: Disco (Discussion of Cost) Provider Companion Intervention

INTERVENTIONS:
Behavioral: Disco (Discussion of Cost) Provider Companion Intervention — A communication intervention for providers to assess financial toxicity in Cancer patients

SUMMARY:
The overall goal of this research program is to address financial toxicity through the development, testing, and implementation of a multi-level communication intervention. If successful, this intervention could be a companion intervention for Cancer providers in combination with the already in testing DISCO app (Discussions of Cost App) for patients. Participants will:

* complete a baseline survey
* attend two one on one meetings, one as part of the development and the second as part of the pilot testing of the intervention.

DETAILED DESCRIPTION:
20 Wayne State University (WSU)/Karmanos Cancer Institute (KCI) oncology care providers (e.g., medical oncologists, nurses, social workers, APP) who treat patients at the KCI Detroit and Farmington Hills clinics where patients are treated for cancer will be recruited. At least two providers from each discipline who treat various cancer types will be included. The study will be discussed at clinic program meetings and then interested providers will be consented. Providers who consent will agree to 1) complete a baseline survey, and 2) attend two one-on-one meetings, one as a part of the DISCO (Discussion of Cost) Provider development (Aim 1) and the second as a part of the DISCO Provider pilot-testing (Aim 2).

To achieve Aim 1, participants will be asked to complete a survey eliciting their demographic and professional characteristics prior to interviews. Then, during one-on-one interviews, which will be audio recorded and subsequently transcribed, the investigators will present the DISCO Provider wireframes and ask participants to provide feedback on the planned content, organization, and implementation. The Investigators will also present participants with strategies identified from research on how to initiate, respond to, and effectively discuss cost concerns. Investigators will ask participants about ideas for website design and training intervention implementation. Participants will be asked to complete a needs assessment interview about their use of digital support tools.

To achieve Aim 2 and pilot test DISCO Provider, participants will again meet one-on-one with the Investigators. Investigators will ask participants to provide feedback on the acceptability and usability of the working version of DISCO Provider, whether participants think it is useful for training providers to discuss cost, if the strategies suggested will likely be effective, and suggestions for improvement. Meetings will be audio recorded, transcribed, and analyzed using similar methods as those in Aim 1

ELIGIBILITY:
Inclusion Criteria:

* Oncology care providers at Karmanos Cancer Institute (KCI)/Wayne State University(WSU) including medical oncologists, nurses, social workers and advance practice providers who treat cancer patients at KCI Detroit or Farmington Hills clinics

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-12-09 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Acceptability - Qualitative report | Immediately Post Pilot Test
  Success of intervention measured by semi-structured qualitative interview method which addresses acceptability
Usability-Qualitative Report | Immediately post pilot test
  Success of intervention measured by semi-structured qualitative interview method which addresses usability
Usefulness-Qualitative Report | Immediately Post Pilot Test
  Success of intervention measured by semi-structured qualitative interview method which addresses usefulness

CONTACTS AND LOCATIONS:
Overall Officials: Lauren M Hamel, PhD, Principal Investigator — Wayne State University
Locations (1):
- Karmanos Cancer Institute, Detroit, Michigan, United States